CLINICAL TRIAL: NCT01670734
Title: An Open-Label, Pharmacokinetic and Tolerability Study of SAR236553/REGN727 Given as a Single SC Dose in Subjects With Mild and Moderate Hepatic Impairment, and in Matched Subjects With Normal Hepatic Function
Brief Title: Pharmacokinetic and Tolerability of Alirocumab SAR236553 (REGN727) in Patients With Hepatic Impairment and in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: POP12671; 2012-002292-33; U1111-1129-0248 (Other: UTN)
Record Dates: First submitted 2012-08-16; First posted 2012-08-22 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- alirocumab SAR236553 (REGN727) - mild hepatic function (Experimental): Injection through subcutaneous (SC) administration in patients with mild hepatic function
  Interventions: Drug: alirocumab SAR236553 (REGN727)
- alirocumab SAR236553 (REGN727) - moderate hepatic function (Experimental): Injection through subcutaneous (SC) administration in patients with moderate hepatic function
  Interventions: Drug: alirocumab SAR236553 (REGN727)
- alirocumab SAR236553 (REGN727) - normal hepatic function (Experimental): Injection through subcutaneous (SC) administration in patients with normal hepatic function
  Interventions: Drug: alirocumab SAR236553 (REGN727)

INTERVENTIONS:
Drug: alirocumab SAR236553 (REGN727) — alirocumab SAR236553 (REGN727) is a fully human monoclonal antibody that binds PCSK9 (proprotein convertase subtilisin/kexin type 9)
  Pharmaceutical form:Solution for injection Route of administration: subcutaneous

SUMMARY:
Primary Objective:

Study the effect of mild or moderate hepatic impairment on the pharmacokinetics of alirocumab SAR236553 (REGN727).

Secondary Objectives:

* Assess the safety and tolerability of alirocumab SAR236553 (REGN727) in patients with mild and moderate hepatic impairment and in matched subjects with normal hepatic function.
* Assess the pharmacodynamic profile of alirocumab SAR236553 (REGN727) in patients with hepatic impairment and in matched subjects with normal hepatic function.

DETAILED DESCRIPTION:
Total duration of the study per subject (excluding screening) is about 12 weeks.

ELIGIBILITY:
Inclusion criteria :

* Male or female, between 18 to 75 years of age, inclusive.
* Patients with mild and moderate hepatic impairment based on Child-Pugh score and stable chronic liver disease.
* Healthy subjects with normal hepatic function.

Exclusion criteria:

* Patients with acute hepatitis, hepatic encephalopathy grade 2, 3, and 4.
* Patients with history or presence of uncontrolled clinically relevant illness.
* Healthy subjects with history or presence of clinically relevant illness.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Assessment of serum concentrations of alirocumab SAR236553 (REGN727) | Up to 12 weeks

SECONDARY OUTCOMES:
Assessment of PK parameter - terminal elimination half-life (t1/2z) [ | Up to 12 weeks
Assessment of PK parameter - apparent total body clearance (CL/F) | Up to 12 weeks
Assessment of PK parameter - Distribution volume at the steady-state (Vss/F) | Up to 12 weeks
Assessment of PK parameter - time to maximum concentration (tmax) | Up to 12 weeks
Assessment of PK parameter - Mean Residence Time (MRT [area]) | Up to 12 weeks
Pharmacodynamics: Change in LDL-C from baseline | Up to 12 weeks
Number of participants with Adverse Events | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Investigational Site Number 250001, Rennes, France
- Investigational Site Number 498001, Chisinau, Moldova